CLINICAL TRIAL: NCT05748314
Title: Marfan Syndrome: the Impact on the Quality of Life, Phenotypic Manifestations on Self-image and Self-management Skills, as an Index of Adaptation to the Disease in Pediatric Patients
Brief Title: Marfan Syndrome and Quality of Life of Pediatric Patients
Acronym: MarfanPed
Status: Active, not recruiting | Type: Observational
Sponsor: IRCCS Policlinico S. Donato (Other)
Responsible Party: Principal Investigator, Alessandro Pini, Principal Investigator, IRCCS Policlinico S. Donato
Other Study IDs: MarfanPed
Record Dates: First submitted 2023-01-26; First posted 2023-02-28 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Rare Diseases; Pediatric Disorder
Keywords: Quality of Life; Self-identification; Self-care
MeSH Terms: conditions — Rare Diseases | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Questionnaire — KINDL-R; Morisky Medication Adherence Scale;

SUMMARY:
The goal of this observational study is to learn about the impact of Marfan syndrome (MFS) in paediatric affected subjects. the main questions it aims to answer are:

* The assessment of quality of life in MFS Italian patients;
* The impact of phenotypic manifestations on self-image and self-management skills;
* Stratify patients according to the need of psychological support. Participants will take part in the study by completing four self-report questionnaires.

DETAILED DESCRIPTION:
In literature, adolescents with MFS experience difficulty in connecting with peers, and are convinced that they would have been more physically attractive without the disease. Additionally, due to physical activity restrictions and orthopedic limitations, these patients reported having difficulty adjusting and participating in educational events.

Data from present study will be able to support clinicians in identifying patients who need psychological support (through parental counseling interviews) aimed at increasing compliance with treatments and adaptation to the disease.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent;
* MFS diagnosis according to Revised Ghent criteria (2010);

Exclusion Criteria:

* Known cognitive deficits

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Subjects with clinical and/or genetic diagnosis od MFS currently in follow up at Cardiovascular Genetic Centre, IRCCS Policlinico San Donato
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2023-01-09 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Psychological counseling | 12 months
  Questionnaire to assess psychological support is KINDL-R (Quality of life);
Psychological counseling | 12 months
  Questionnaire to assess psychological support is Multidimensional Self Concept Scale (MSCS)
Psychological counseling | 12 months
  Questionnaire to assess psychological support is Morisky Medication Adherence Scale

CONTACTS AND LOCATIONS:
Overall Officials: Alessandro Pini, MD, Principal Investigator — Cardiovascular-Gentic Centre, IRCCS Policlinico San Donato
Locations (1):
- IRCCS Policlinico San Donato, San Donato Milanese, Lombardy, Italy

IPD SHARING:
Plan to Share IPD: Undecided